CLINICAL TRIAL: NCT05731518
Title: A Phase Ib/II , Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Effects of SC0245 in Combination With Irinotecan in Patients With ES-SCLC
Brief Title: SC0245 and Irinotecan in Treating Patients With Relapsed Extensive-Stage Small Cell Lung Cancer (ES-SCLC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC0245-102
Record Dates: First submitted 2023-01-09; First posted 2023-02-16 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SC0245 and irinotecan combination (Experimental): SC0245 and irinotecan combination are administered one cycle that is consisted of 28 days until disease progression or death or loss of follow-up or withdrawal.
  Interventions: Drug: SC0245; Drug: Irinotecan

INTERVENTIONS:
Drug: SC0245 — SC0245 Quaque Die(QD) administered with a 3-day on and 4-day off schedule in Day 1 Day8 and Day 15 of each cycle. One cycle is consisted of 28 days.
  Other Names: SC0245 tablet
Drug: Irinotecan — Irinotecan 80mg/m^2 via IV administered for every 4 weeks (fixed dosing) in Day 1 Day8 and Day 15 of each cycle. One cycle is consisted of 28 days.
  Other Names: Irinotecan hydrochloride injection

SUMMARY:
This study is a single arm, multi-center, open label phase Ib/II study of SC0245 and Irinotecan combination therapy in subjects with extensive-stage small cell lung cancer (ES-SCLC) as a second therapy. This study will have three parts, phase 1 dose escalation (Part 1), phase 1 dose expansion (Part 2), and phase 2 combination therapy (Part 3).

DETAILED DESCRIPTION:
This study will have three parts, phase 1 dose escalation (Part 1), phase 1 dose expansion (Part 2)， and phase 2 combination therapy (Part 3).

Subjects will receive SC0245 and Irinotecan combination therapy. The study is composed of 67 subjects.

Irinotecan 80mg/m2 via IV administered for every 4 weeks (fixed dosing) in Day 1 Day8 and Day 15 of each cycle, and SC0245 administered with a 3-day on and 4-day off schedule in Day 1 Day8 and Day 15 of each cycle. One cycle is consisted of 28 days.

Study treatment will be continued until objective disease progression (unless other criteria for treatment discontinuation are met). Tumor evaluation using CT or MRI by RECIST 1.1 every 8weeks(±1week) until objective disease progression. RECIST 1.1 scans will be analyzed by the investigator on site. If a subject discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

Primary Objective:

Part 1 (phase 1 dose escalation): To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of SC0245 in combination with irinotecan in patients with advanced solid tumors.

Part 2 (phase 1 dose expansion): To evaluate the safety and tolerability of SC0245 in combination with irinotecan in patients with relapsed extensive-stage small cell lung cancer (ES-SCLC).

Part 3(phase 2 combination therapy): To evaluate the preliminary anti-tumor activity of SC0245 in combination with irinotecan in patients with relapsed extensive-stage small cell lung cancer (ES-SCLC).

Secondary Objective:

Part 1 (phase 1 dose escalation): To characterize the PK profile and the preliminary anti-tumor activity.

Part 2 (phase 1 dose expansion): To characterize the PK profile, safety and tolerability and the preliminary anti-tumor activity in patients with relapsed extensive-stage small cell lung cancer (ES-SCLC).

Part 3(phase 2 combination therapy): To characterize the safety and tolerability and the preliminary anti-tumor activity in patients with relapsed extensive-stage small cell lung cancer (ES-SCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumor.
2. Phase 1b dose-escalation stage: patients with advanced solid tumors, who have received standard treatment, for who no standard treatment exists, who are not suitable for standard treatment at the current situation, or who could not tolerate standard treatment.

   Phase 1b dose-expansion stage and phase 2: patients with ES-SCLC who have received first-line platinum-based regimen chemotherapy with or without immunotherapy or intolerance to such therapy.
3. Measurable lesions according to RECIST version 1.1 (only applicable for phase 1b dose-expansion and Phase 2).
4. Male or non-pregnant, non-lactating female patients age ≥18 years on day of signing the informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
6. Life expectancy ≥ 3 months.
7. Adequate organ function .
8. Females of child-bearing potential (nonlactating) must have a negative blood pregnancy test within 7 days before enrollment, and must agree to use a medically effective contraception from the time they provided the informed consent until at least 6 months (or at least 180 days) after the last dose of study drug, unless surgical sterilization or menopause for more than 1 year. Patients who are sexually active men with a female partner of child-bearing potential must agree to use adequate contraception from the time they provided informed consent until at least 6 months after the last dose.
9. Subjects voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Received chemotherapy within 3 weeks before first dose of study drug (6 weeks for nitrosoureas or mitomycin C)
2. Received wide field radiotherapy within 4 weeks before first dose of study drug (previous palliative radiation therapy for metastatic disease is permitted if it has been completed at least 1 week before first dose of study drug and related toxicity has recovered to ≤ grade 1)
3. Received any monoclonal antibody, radioimmunoconjugate or antibody-drug conjugates (ADC) within 5 half-lives or 4 weeks (whichever is shorter) before first dose.
4. Received any other type of anti-tumor therapy including other investigational drugs or treatments not listed above within 4 weeks before first dose of study drug.
5. Had major organ surgery, except diagnostic biopsy, or significant trauma within 4 weeks, or not fully recovered from surgery within 4 weeks before first dose of study drug.
6. Received traditional Chinese herbal medicines with anti-tumor indications within 2 weeks before first dose of study drug.
7. Previously received any Ataxia-Telangiectasia and Rad3 Related（ATR）inhibitor.
8. Continuous toxicities due to prior treatments that do not recover to ≤ Grade 1 severity per NCI CTCAE v5.0 except for clinically non-significant events judged by the Investigator (e.g., alopecia, grade 2 peripheral neurotoxicity, stable hypothyroidism with hormone replacement therapy, etc.)
9. Allergy to any component of the SC0245 tablets and irinotecan injection or who meet contraindications to irinotecan. In addition, the prohibited concomitant drugs in irinotecan label should be avoided.
10. Crigler-Najjar syndrome (Type I and II) or UGT1A1 mutation that increases irinotecan toxicity (Gilbert's syndrome).
11. Central nervous system (CNS) metastases meeting any of the following condition:

    * Presence of new or progressive lesions in brain by imaging within 4 weeks prior to first dose of study drug
    * Presence of symptoms of CNS metastasis
    * Received corticosteroids, radiotherapy, or dehydration drugs within 1 week to control symptoms of CNS metastasis (except for patients who completed radiotherapy for brain metastases, no use of cortisol and dehydration drugs without neurologic symptoms for more than 1 week, and brain metastases are in a stable state or have shrinkage during follow-up visit at least 2 weeks later, which need to be confirmed before first dose of study drug)
    * Carcinomatous meningitis
    * Brain stem (midbrain, pons, medulla oblongata) and spinal cord metastases
12. Active infections that require systematic treatment
13. Severe cardiovascular disorder, who meet any of the following conditions:

    * corrected QT interval(QTc)> 470 ms
    * Severe cardiac rhythm or conduction abnormalities, including but not limited to complete left bundle branch block, atrioventricular block of degree II or above, rapid ventricular tachycardia (including frequent premature ventricular contractions), torsades de pointes.
    * Any risk factors that increase the prolongation of the QTc interval, such as uncorrectable hypokalemia, genetic long QT syndrome, taking medications that prolong the QTc interval (mainly antiarrhythmic drugs of Class Ia, Ic, or III)
    * Congestive heart failure (New York Heart Association Class≥3), or a left ventricular ejection fraction of less than 50%
    * Clinically uncontrolled hypertension, defined as systolic blood pressure (SBP) ≥ 160 mmHg and diastolic blood pressure (DBP) ≥ 100 mmHg after medication.
    * Acute coronary syndrome, aortic dissection, myocardial infarction, unstable angina pectoris, cerebrovascular accident, or other Grade 3 or higher cardiovascular or cerebrovascular event within 6 months prior to the first dose
14. Major gastrointestinal surgery, or malabsorption syndrome, or are unable to swallow tablets that may impair the absorption of SC0245 tablets, or other active diseases or pathological conditions that may impact absorption, distribution, metabolism, excretion of SC0245 (such as uncontrollable nausea, vomiting, diarrhea, intestinal obstruction) as judged by the Investigator within 4 weeks before first dose of study drug.
15. Tertiary-interstitial effusion (e.g., pericardial, pleural, and peritoneal effusion) requiring repeated drainage or other treatments, but still could not be controlled within two weeks before first dose of study drug and are judged unsuitable to participate in the study by the Investigator.
16. Patients with other known malignant diseases. Exceptions: History of curative treatment for malignancy with no recurrence within 5 years; adequately treated non-melanoma skin cancer or lentigo malign; carcinoma in situ adequately treated with no signs of recurrence
17. UGT1A1 mutation.
18. Patients with underlying medical conditions (including laboratory abnormalities), alcohol or drug abuse or dependence that may affect study drug administration or the interpretation of drug toxicity or adverse events (AEs), or result in poor compliance, and are judged unsuitable to participate in the study by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Part 1 (phase 1 dose escalation):Maximum tolerated dose (MTD), and recommended phase 2 dose (RP2D) of SC0245 and irinotecan | Up to 28 days
  MTD Will be defined as the highest dose level at which =< 30% patients experience dose limiting toxicity. Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optional therapeutic intervention, meets protocol-defined criteria. The RP2D will be determined based on MTD and the feasibility of the administration.
Part 2 (phase 1 dose expansion):Safety and tolerability in terms of adverse events | From the first dose of study treatment until 30 days after the last dose, up to approximately 24 months
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters.
Part 3(phase 2 combination therapy):Objective response rate (ORR) | Up to 24 months.
  Defined as the percentage of participants having a CR or PR based on investigator assessment per RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) Based on RECIST v1.1 | Assessed every 8 weeks, up to 24 months.
  Defined as the percentage of participants having CR, PR, or stable disease (SD) based on investigator assessment per RECIST v1.1.
Duration of Response (DoR) Based on RECIST v1.1 | Assessed every 8 weeks, up to 24 months.
  Defined as the time from the earliest date of disease response (CR or PR) until earliest date of disease progression or death due to any cause.
Progression-free Survival (PFS) Based on RECIST v1.1 | Assessed every 8 weeks, up to 24 months.
  Defined as the time from the start of combination therapy until the earliest date of disease progression or death due to any cause.
Overall Survival (OS) | At 1 year and 2 years.
  Defined as the time from the start of combination therapy until death due to any cause.
Incidence of adverse events of SC0245 and irinotecan | From the first dose of study treatment until 30 days after the last dose, up to approximately 24 months
  Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. A toxicity will be considered to be an adverse event that is possibly, probably or definitely related to treatment. The maximum grade of toxicity for each category of interest will be recorded for each patient, and the summary results will be tabulated by category, grade, and dose level. Serious (>= grade 3) toxicities will be described on a patient-by-patient basis and will include any relevant baseline data.
Maximum observed blood concentration (Cmax) of SC0245 | Pre-dose up to approximately 6 months
  Defined as assessments for measuring maximum blood concentration of SC0245
AUC Area under the Plasma Concentration versus Time Curve (AUC) of SC0245 | Pre-dose up to approximately 6 months
  Defined as assessments for evaluating the Area Under the Concentration-Time Curve (AUC)
Elimination half-life (t1/2) of SC0245 | Pre-dose up to approximately 6 months
  Defined as the time required for half of the drug SC0245 to be eliminated from the blood.

CONTACTS AND LOCATIONS:
Overall Officials: SHUN LU, Prof, Study Chair — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China